CLINICAL TRIAL: NCT07274631
Title: A Cohort for Inflammatory Respiratory Diseases: From Phenotyping to Personalised Medicine
Acronym: PALMIRE
Status: Not yet recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PL25060*
Record Dates: First submitted 2025-06-10; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Bronchiectasis; Cystic Fibrosis; Primary Ciliary Dyskinesia
Keywords: Chronic obstructive pulmonary disease; Asthma; Bronchiectasis; Cystic fibrosis; Primary ciliary dyskinesia; Airway microbiota; Airway epithelium; Remodeling; Exposome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Bronchiectasis; Cystic Fibrosis; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non applicable — Non applicable

SUMMARY:
Chronic inflammatory pulmonary diseases, including asthma, chronic obstructive pulmonary disease (COPD), bronchiectasis, cystic fibrosis (CF), primary ciliary dyskinesia (PCD) and interstitial lung diseases (ILD) are characterised by lung inflammation and remodelling. Clinical, functional, microbiological, biological, pathological and prognostic features are highly variable and heterogeneous. Several phenotypes have been described within the same pathology, as similar phenotypic traits between different pathologies, or the coexistence of components of several diagnoses in the same patient, suggesting shared underlying mechanisms that could represent new therapeutic targets, beyond the initial medical diagnosis.

The objectives of this prospective study are to analyze the phenotypic characteristics (clinical, demographic, biological, morphological, pathological, and microbiological characteristics) together with respiratory exposures and underlying mechanisms involving airway epithelium and inflammation processes in a cohort of patients diagnosed with asthma, COPD, bronchiectasis, CF, PCD and ILD.

DETAILED DESCRIPTION:
The cohort for inflammatory respiratory diseases: from phenotyping to personalised medicine (The PALMIRE project) is a monocentric study conducted at the University Hospital of Reims, France.

Study Population :

Adult patients (>18 year-old) followed at the University Hospital of Reims and diagnosed with asthma, COPD, bronchiectasis, CF, PCD, and IPF will be considered for inclusion. Patients will sign an informed consent for inclusion. Exclusion criteria include "subjects protected by the law" as required by the French authorities. Control patients with no respiratory diseases after clinical and pulmonary function tests assessment will also be included. The expected number of patients included is 470 (Asthma, n=100; COPD, n=150; bronchiectasis, n=50; CF, n=60; PCD, n=30; ILD, n=30; controls, n=50). Inclusion will be conducted for 60 months from July 2025 to July 2030.

Study Procedures:

For all asthma, COPD, bronchiectasis, CF, PCD, and IPF patients included, data will be registered at inclusion, and at follow-up visits for 10 years. Patients will be followed-up as usual care with no specific therapeutic intervention. For control patients, data will be registered at inclusion with no follow-up.

The recorded data will include demographics, history of respiratory disease and comorbidities, respiratory symptoms, results of lung function tests and CT-scan, microbiological and pathological features of respiratory sampling when performed.

Data Analysis:

Data will be registered in a centralized anonymized database. The characteristics of the patients will be described as mean and standard deviation for quantitative data and as number and percentages for qualitative data. Comparisons and associations between groups and variables will be analyzed by Student, Wilcoxon, Chi2, Fischer exact, and Spearman tests as applicable. A p<0.05 will be considered as significant. Multivariate and longitudinal statistical models will be used to identify clusters of patients with shared endotypes. Machine learning approaches will be employed to integrate multi-omic data and generate predictive models for disease trajectories and treatment responses.

Significance:

This study should help better understand the pathogenesis and heterogeneity of chronic respiratory diseases by integrating the analysis of phenotypic and endotypic characteristics of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Follow-up for one of the following conditions: asthma, COPD, bronchiectasis (DDB), cystic fibrosis (CF), primary ciliary dyskinesia (PCD), or interstitial lung diseases (ILD)
* Healthy volunteers (controls)

Exclusion Criteria:

* Subjects protected by law (e.g., legal incapacity)
* Any condition preventing informed consent or participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) followed for chronic inflammatory respiratory diseases (asthma, COPD, bronchiectasis, cystic fibrosis, primary ciliary dyskinesia, or interstitial lung diseases) at the Respiratory Medicine Department of CHU Reims. Healthy control subjects without diagnosed respiratory disease will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
pheno-endotypes of inflammatory respiratory disease | Baseline
  Number of subjects in each of the identified pheno-endotypes of inflammatory respiratory disease

SECONDARY OUTCOMES:
Forced expiratory volume in one second ( FEV1) | 10 years
Forced Vital Capacity ( FVC ) | 10 years
Total Lung Capacity (TLC) | 10 years
Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) | 10 years
6 minutes walking distance | 10 years
Modified Medical Research Council Dyspnea Scale (mMRC dyspnea score) | 10 years
Asthma Control Test (ACT questionnaire score) | 10 years
Cough and Sputum Assessment Questionnaire (CASA-Q questionnaire score) | 10 years
Asthma Quality of Life Questionnaire (AQLQ score) | 10 years
St George's Respiratory Questionnaire (SGRQ score) | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided